CLINICAL TRIAL: NCT05035264
Title: Head Position for Laryngeal Mask Air Leak and Performance in Paediatric Patients (Neutral, Sniffing and Beyond Sniffing Position): Prospective Randomized Trial
Brief Title: Head Position for Laryngeal Mask Air Leak and Performance in Paediatric Patients (Neutral, Sniffing and Beyond Sniffing Position)
Acronym: SNIFFLMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KDAR SNIFF LMA
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Airway Management
Keywords: Supraglottic Airway Devices; Laryngeal mask airway; Head position; Paediatric patient

STUDY DESIGN:
Intervention Model Description: Paediatric patients (between 2-18 years) undergoing elective airway management without predicted/confirmed difficult airway with the laryngeal mask airway after anaesthesia induction
Who Masked: Participant
Masking Description: Under general anaesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neutral head position (Active Comparator): Laryngeal mask will be inserted after anaesthesia induction in neutral head position
  Interventions: Device: Laryngeal mask insertion
- Sniffing position (Active Comparator): Laryngeal mask will be inserted after anaesthesia induction in sniffing head position
  Interventions: Device: Laryngeal mask insertion
- Beyond sniffing position (Experimental): Laryngeal mask will be inserted after anaesthesia induction in sniffing head position
  Interventions: Device: Laryngeal mask insertion

INTERVENTIONS:
Device: Laryngeal mask insertion — Laryngeal mask insertion in neutral position
Device: Laryngeal mask insertion — Laryngeal mask insertion in sniffing position
Device: Laryngeal mask insertion — Laryngeal mask insertion in beyond sniffing position

SUMMARY:
The correct head position for airway management is considered as a mainstay of good clinical practice. The recommended head position for all patients is the horizontal position of the head with in tragus-to- sternal notch in line alignment. This could be achieved in infant (under two years) supporting the shoulder, neutral head positioning in children between 2-8 (12) years and with so called "sniffing position" (SP) in patients over 12 year by supporting the head (i.e. with pillow) to reach the proper alignment (tragus to sternal notch). Although, this could be considered as gold standard, there are currently insufficient high quality evidence-based data to confirm the association between the better laryngeal view during the direct laryngoscopy and tragus-to-sternal notch position. Recently, "beyond sniffing" position was described as further head elevation (compared to sniffing position) in adult patients. Beyond sniffing position was associated with superior laryngeal inlet visualization compared to standard sniffing position in common elective adult airway management (patients with suspected or confirmed difficult airway was excluded). The hypothesis of SNIFF LM trial is that the sniffing position or even beyond sniffing position could be associated with superior laryngeal mask performance (lower incidence of air leak, LM easier introduction) compared neutral position in paediatric patients undergoing elective paediatric anaesthesia

DETAILED DESCRIPTION:
Paediatric patients (between 2-18 years) undergoing elective airway management without predicted/confirmed difficult airway will be eligible for inclusion. The patients will be screened for eligibility during the preanaesthesia visit in anaesthesiology examination room. After informed consent the patients will be randomized into 3 groups (according to the induction head position) - neutral head position (without head elevation, head supported with the hollow foam circle to prevent side head movement), sniffing position (head support with inflatable pillow the reach the horizontal in-line alignment of tragus-to-sternal notch line) and beyond sniffing position (further 25% increase of head support compared to sniffing position). The randomization will be performed by the Institute of Biostatistics and Analysis in form of sealed envelopes. The group allocation will be 1:1:1. After fulfilling the inclusion criteria and obtaining the informed consent the patient will be randomized into 3 groups. Before anaesthesia induction the head of the patient will be positioned into the predefined position according to the results of randomization. The anaesthesia induction could be performer either inhalation or intravenous route. After anaesthesia induction, the laryngeal mask will be inserted in the selected position. After laryngeal mask insertion, stabilisation of vital signs and of anaesthesia depth, the measurement will be intiated within 5 minutes. After one minute of ventilation 3 leak volumes (inspiration - expiration tidal volume) together with the peak airway pressure (3 measurements) will be recorded (the mean volume and mean pressure will be analyzed). Patient´s head will be repositioned into the 2nd position and after one minute of ventilation leak volume and airway pressure will be recorded as previously described, after measurement, the head position will be repositioned into the 3rd positon and the measurement will be repeated. The incidence of 1st insertion attempt failure rate, incidence of laryngeal mask failure rate, incidence of the need for reposition will be recorded together with the incidence of airway related complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-19 years
* Informed consent
* Elective airway management
* laryngeal mask for airway management

Exclusion Criteria:

* Outside the age limits
* Decline to participate
* Predicted or confirmed difficult airway
* Cervical spine injury
* limited access to head of the patient after anaesthesia induction (for the measuement purposes)
* Intubation

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
leak volume in 3 different head position in every patient (1st position will be randomized) | 1 minute mechanical ventilation in predefined head position
  leak volume in 3 different head position in every patient (1st position will be randomized) defined by the average leak obtained from 3 measurements in selected position

SECONDARY OUTCOMES:
Leak pressure in 3 different head position in every patient (1st position will be randomized) | 1 minute mechanical ventilation in predefined head position
  Leak pressure in 3 different head position in every patient (1st position will be randomized) defined by the first audible leak during stepwise increasing inspiratory pressure
incidence of failed 1st attempt insertion rate | anaesthesia induction
  incidence of failed 1st attempt insertion rate
incidence of overall laryngeal mask failure | anaesthesia induction
  incidence of overall laryngeal mask failure
incidence of the need for head reposition to obtain better airway seal in the 3 randomized head positions. | Intraoperatively
  incidence of the need for head reposition to obtain better airway seal in the 3 randomized head positions
Incidence of airway related complication | From anaesthesia induction until dismission from postanaesthesia care unit
  Incidence of airway related complication -regurgitation/aspiration, desaturation, oesophageal intubation, laryngeal/airway injury incidence

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided